CLINICAL TRIAL: NCT06787014
Title: Resection of the Primary Tumor vs. Systemic Treatment Alone for Patients With Small Intestinal Neuroendocrine Tumors and Unresectable Metastases: a Retrospective, Europe-wide, Pooled Cohort Study (ENETS-SurgSmInt)
Brief Title: Resection of the Primary Tumor vs. Systemic Treatment Alone for Patients With Small Intestinal Neuroendocrine Tumors and Unresectable Metastases: a Europe-wide Study
Acronym: ENETSSurgSmInt
Status: Not yet recruiting | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: ENETSSurgSmInt
Record Dates: First submitted 2025-01-07; First posted 2025-01-22 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Neuroendocrine (NE) Tumors; Metastasis; Bowel Obstruction
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis; Intestinal Obstruction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Histopathological review: The patients will be grouped according to whether a primary tumor resection within 6 months after initial diagnosis was performed (yes vs. no).
  Interventions: Other: Histopathological review

INTERVENTIONS:
Other: Histopathological review — Histopathological review

SUMMARY:
When possible, surgery to completely remove small intestinal neuroendocrine tumors (siNETs) is always recommended. However, in cases where the tumor has spread and cannot be cured completely, it is unclear whether a surgical removal of the primary tumor only is reasonable. In this situation, current guidelines from the European Neuroendocrine Tumor Society (ENETS) recommend surgery only for patients who have symptoms like intestinal blockage or bleeding, or are at risk of such complications. For patients without symptoms, it is still unclear whether removing the main tumor improves overall outcomes and prevents future problems.

Studies evaluating this type of surgery on survival show conflicting results. These studies often do not separate patients with symptoms from those without, and they overlook other important factors like the amount of cancer in the liver and nearby tissues. Due to these uncertainties, the rarity of siNETs and many factors that can affect outcomes, like age, overall health, or other current treatments, conducting a high-quality study to answer this question is challenging. To address this, the present Europe-wide study is being planned.

This study aims to determine if resecting the main tumor improves the 10-year overall survival and reduces risks like intestinal blockages or blood flow issues compared to no surgery in patients without symptoms. The study will also assess other outcomes, such as how long patients stay free from disease progression, the risks of surgery, and prognostic factors for long-term survival. This international collaboration among neuroendocrine tumor referral centers will provide robust evidence to guide clinical practice and update treatment guidelines for siNETs.

ELIGIBILITY:
Inclusion Criteria:

- All patients with siNET and non-curative metastatic disease between 01.01.2005 and 31.12.2019 will be included.

Exclusion Criteria:

- All patients with siNET G3, resectable metastatic disease and/or non-resectable primary tumor at initial diagnosis will be excluded. Furthermore, symptomatic patients (small intestinal obstruction, bleeding) or when imaging suggests that obstruction will probably occur (bowel dilatation, mesenteric fibrosis) at initial diagnosis will be excluded. Patients with diarrhea, flushing, or abdominal pain will not be excluded.

Patients with a documented rejection for a further use of their data for scientific purposes will also be excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The investigators will include all patients with siNET and non-curative metastatic disease between 01.01.2005 and 31.12.2019.
Sampling Method: Non-Probability Sample
Enrollment: 3200 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2025-07-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
To evaluate the 10-year overall survival of non-curative metastatic siNET with or without primary tumor resection at initial diagnosis in asymptomatic patients. | 10 years follow-up
  For the survival analysis, Kaplan-Meier method will be used to estimate overall survival at 10 years for patients with and without primary tumor resection.

SECONDARY OUTCOMES:
To evaluate the progression-free survival of non-curative metastatic siNET with or without primary tumor resection at initial diagnosis in asymptomatic patients. | 10 years follow-up
  For the survival analysis, Kaplan-Meier method will be used to estimate overall survival at 10 years for patients with and without primary tumor resection.
To examine the risk of small intestinal obstruction with or without palliative primary tumor resection | 10 years follow-up
  To account for additional established prognostic information, univariable and multivariable Cox proportional hazards regression will be used.
To examine the risk of small intestinal hypoperfusion with or without palliative primary tumor resection | 10 years follow-up
  To account for additional established prognostic information, univariable and multivariable Cox proportional hazards regression will be used.
To evaluate the morbidity of palliative primary tumor resection | 10 years follow-up
  To account for additional established prognostic information, univariable and multivariable Cox proportional hazards regression will be used.
To evaluate the mortality of palliative primary tumor resection | 10 years follow-up
  To account for additional established prognostic information, univariable and multivariable Cox proportional hazards regression will be used.
To assess prognostic factors for long-term survival | 10 years follow-up
  The following prognostic information will be taken into account: age, sex, ECOG, presence of second malignancy, and adjusted for characteristics of the siNET (Ki-67 index, number of siNETs, lymph node metastases, TBS, extrahepatic metastases, CgA level, 5-HIAA level, carcinoid heart disease, and use of other treatments), with results presented as adjusted hazard ratios (HRs) and 95% CI.

CONTACTS AND LOCATIONS:
Overall Officials: Reto Kaderli, Principal Investigator — Insel Gruppe AG, University Hospital Bern
Locations (1):
- UHI Berne, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No